CLINICAL TRIAL: NCT02167698
Title: A Parallel-arm, Single Blind Randomised Controlled Trial Comparing 'AIRWAY PRESSURE RELEASE VENTILATION' and 'LOW-TIDAL VOLUME VENTILATION' in Children With Acute Respiratory Distress Syndrome
Brief Title: Trial of an Alternate Mode of Providing Artificial Breaths to Children With Very Severe Pneumonia
Acronym: APRiCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Increased mortality in the intervention arm at 50% enrolment
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Saptharishi L G, MBBS, MD, DM (Pediatric Critical Care) Senior Resident, Division of Pediatric Critical care, Dept. of Pediatrics, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTRI/2014/06/004677; CTRI/2014/06/004677 (Registry Identifier: Clinical Trials Registry of India)
Record Dates: First submitted 2014-06-16; First posted 2014-06-19 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: Pediatric acute respiratory distress syndrome; Mechanical ventilation; Airway pressure release ventilation; Conventional low-tidal volume ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Continuous Positive Airway Pressure; Methylprednisolone; Interleukin-6; Interleukin-8

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Airway pressure release ventilation arm (Experimental): This group of children would be ventilated using the Airway pressure release ventilation (APRV) mode.
  Restrictive fluid therapy, protocolized sedo-analgesia titration, steroid therapy, protocolized supportive care, protocolized early enteral nutrition would be provided to both the groups. Biomarkers would be measured in both groups.
  Interventions: Device: Airway Pressure Release Ventilation (APRV); Drug: Methylprednisolone; Other: Restrictive fluid therapy; Drug: sedo-analgesia titration; Other: Protocolized early enteral nutrition; Other: Protocolized supportive care; Other: Biomarker Assay
- Low-tidal volume ventilation arm (Active Comparator): Low-tidal volume ventilation using pressure-regulated volume control mode with target tidal volume of 6 ml/kg or less and other lung-protective strategies. Restrictive fluid therapy, protocolized sedo-analgesia titration, steroid therapy, protocolized supportive care, protocolized early enteral nutrition would be provided to both the groups. Biomarkers would be measured in both groups
  Interventions: Other: Low-tidal volume ventilation; Drug: Methylprednisolone; Other: Restrictive fluid therapy; Drug: sedo-analgesia titration; Other: Protocolized early enteral nutrition; Other: Protocolized supportive care; Other: Biomarker Assay

INTERVENTIONS:
Device: Airway Pressure Release Ventilation (APRV) — This is a newer mode of ventilation that has been hypothesized to be equivalent or even superior to the conventional low-tidal volume mode of ventilation
  Other Names: BiLevel; BiPAP
  Arms: Airway pressure release ventilation arm
Other: Low-tidal volume ventilation — This mode of ventilation is the standard of care worldwide for ventilating children with ARDS.
  Other Names: Lung-protective ventilation
  Arms: Low-tidal volume ventilation arm
Drug: Methylprednisolone — Children with primary ARDS presenting within the first 14 days would receive IV low dose Methylprednisolone infusion.
Other: Restrictive fluid therapy — Fluid & hemodynamics would be titrated as per pre-designed decision-making protocols
Drug: sedo-analgesia titration
Other: Protocolized early enteral nutrition — Early enteral nutrition and attempt to meet calorie-protein goals
Other: Protocolized supportive care — Eye care, chlorhexidine mouth wash Q6 hourly, Strict aseptic precautions prior to any procedures, Skin care & bed sore prevention, Adequate pulmonary toileting and chest physiotherapy, frequent position changes, limb physiotherapy, family-centered care
Other: Biomarker Assay — Biomarker Assay for patients in both arms
  Other Names: Interleukin 6, Interleukin 8, Angiopoeitin-2, soluble-ICAM-1

SUMMARY:
This study attempts to study a new ventilation mode in children with Acute respiratory distress syndrome (ARDS). Despite decades of research, no intervention has brought about a significant decrease in ARDS mortality. Moreover, most of the studies are adult-based and have been extrapolated to children. Airway pressure release ventilation (APRV) mode is hypothesized to be superior in terms of lower need for sedation, shorter duration of mechanical ventilation, etc. It is unique and the first worldwide randomized controlled trial on APRV mode in children.

We plan to recruit a minimum of 50 children aged (1 month-12 years) in each group. The study is to be conducted at the Post-Graduate Institute of Medical Education and Research (PGIMER), Chandigarh between March 2014 to March 2016. This trial would recruit children with respiratory failure and early ARDS and, randomize them to receive either conventional ventilation or the APRV mode. Rest of the supportive care has also been protocolized so that both groups receive treatment as per the existing best practices in every aspect. The primary outcome being studied is the number of ventilator-free days. The secondary outcomes include length of PICU stay, hospital stay, organ-failure free days, 28 day & 3 month survival, biomarkers of lung injury (IL-6, IL-8, Angiopoeitin-2, soluble-ICAM-1, etc), functional status, Pulmonary function tests, etc. Funding request would be sent to the Indian Council of Medical Research, New Delhi, India.

Assessing lung biomarkers like Interleukin-6 would assess the role of different modes of ventilation in acting as triggers for multi-organ dysfunction as well as for worsening lung injury. This pathbreaking research is likely to open up new avenues upon completion.

DETAILED DESCRIPTION:
Study setting:

15-bedded pediatric intensive care unit (PICU) of a multi-specialty, tertiary referral and teaching hospital- the Advanced Pediatrics Centre (APC) in Post-Graduate Institute of Medical Education and Research (PGIMER), Chandigarh, India Study period Recruitment: January 2014 to December 2016 Data Analysis: Jan 2017 to June 2017 Study design An open-labelled, parallel-arm, efficacy/feasibility randomized controlled trial Ethics approval Ethics approval has been obtained from the Institute Ethics Committee. The study has been registered with Clinical Trials Registry - India (CTRI) (ctri.nic.in). Informed consent will be obtained from the parents/legal guardian and the conversation would be recorded using a camera (audio-visual documentation of evidence).

Sample size estimation Assuming alpha error of 5% and power of 80% with non-inferiority limit of 4 days (Standard deviation of VFDs being 8.2 days in the conventional low tidal volume ventilation group in pilot trial), sample size was calculated to be 52 per group. As this is a safety and feasibility trial, an interim analysis would be done at 50% enrolment.

Enrolment Parents or legal guardians of children who satisfy the above eligibility criteria will be invited by the investigator to participate in the study. Parents are free not to participate, or to withdraw from the study at any point of time. All children, irrespective of their enrollment in the study, will receive standard pediatric intensive care unit (PICU) care as per the unit's existing protocol. An information sheet (in Hindi/ English) furnishing details of the study will be provided to the parents. Given the fact that all these children are sedated and on mechanical ventilation, obtaining assent would not be feasible in this study.

Randomization Sequence generation A computer-generated, unstratified, block randomization with variable block sizes will be performed to determine group allocation. A person not involved in the study will perform the random number allocation and prepare opaque, sealed envelopes containing the allocation.

Concealment allocation Each pre-sealed opaque envelope would be opened only after obtaining a written consent and audio-visual record of the same. As the randomization is done using a variable block size, and prepared by a statistician not directly involved in the study, there would be no way of predicting the random allocation, thus minimizing the risk of allocation bias.

Randomization implementation After parents provide informed consent, randomization would be done within the next one hour and child initiated on appropriate mode of ventilation. The supportive care for both the groups, would be as per the attached supplementary protocols

Intervention protocol:

The Airway pressure release ventilation (APRV) intervention protocol has been designed based on the available APRV literature as of Dec 2013.

Start the child on APRV mode of ventilation with the following settings:

* P HIGH would determine the degree of baseline lung inflation. A rough estimate can be obtained based on the plateau pressure requirements on the conventional mode of ventilation. Perform an inspiratory hold to ascertain the plateau pressures:

  * If P plateau > 30 cm water, set P HIGH at 30 cm water
  * If P plateau < 30 cm water, set P HIGH at or 1-2 cm above the measured P plateau.
* Alternatively, if P plateau cannot be measured, P HIGH can be set according to the following guide:

PaO2/ FiO2 ratio P High < 250 15-20 < 200 20-25 < 150 25-28

After initiating a particular P HIGH, a clinical assessment of lung volume needs to be followed with a chest radiograph to determine the degree of lung inflation (similar to setting of Mean airway pressure in High frequency oscillatory mode of ventilation). The child's P HIGH is adjusted to maintain optimal lung volume, without clinical or radiological evidence of hyperinflation: no signs of decreased cardiac output/ hypotension and/or the level of the diaphragm visible greater than the ninth rib.

* Start at T High of 4 seconds; Titrate T High based on oxygenation status. At least 80 -95% of the total cycle time should be spent in T High.
* Set P Low at Zero cm H2O
* Set T Low so that expiratory flow decreases by 25 % of peak expiratory flow rate (PEFR); usually 0.1-0.8 seconds. The ratio of T-PEFR to PEFR should be targeted near 75%. This entity needs to be titrated every 2-4 hours and may have to be shortened as lung injury advances.
* Set Pressure Support at ZERO
* The number of breaths per minute or number of releases is a function of T High and T Low as depicted below:

Weaning from APRV would also be carried out in a structured, protocolized manner. The following strategies would be adopted:

1. As child's clinical condition and oxygenation index improves, and Fraction of inspired oxygen levels are brought down to 0.6, T HIGH is increased in steps of 0.5-2 seconds till it is 10-12 seconds.
2. P HIGH can be subsequently decreased in steps of 2-3 cm H2O till a value of 12-16 is reached. Decrease in P HIGH can be carried out earlier if features of hyperinflation (clinical/radiological) appear at any point.
3. The goal is to reach pressure levels of 12-16 cm H2O and then switch to Continuous positive airway pressure (CPAP) of 6-8 cm H2O, from which child can be extubated directly to nasal prong CPAP or gradually tapered off CPAP to Endotracheal-T piece and subsequently extubated depending on the overall clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month- 12 years, who are intubated and mechanically ventilated with the following criteria of Acute Respiratory Distress Syndrome:

  1. Acute presentation within 1 week of a known clinical insult or new/ worsening respiratory symptoms
  2. Bilateral opacities on chest imaging - not fully explained by effusions, lobar/lung collapse, or nodules
  3. Respiratory failure is not fully explained by cardiac failure or fluid overload (Echocardiographic assessment to exclude hydrostatic edema)
  4. Impaired oxygenation with PaO2/ FiO2 ratio less than 300 or Oxygenation Index greater than 5.3

Exclusion Criteria:

* Greater than 24 hours since diagnosis of ARDS
* Co-existing raised intra-cranial pressure/ any other condition necessitating use of high dose of sedation (likely to suppress spontaneous breathing)
* Radiologically confirmed air leak prior to randomization - Pneumothorax/ Pulmonary interstitial Emphysema
* Clinical evidence of significant airway obstruction/ severe bronchospasm / reactive airway disease
* Have received mechanical ventilation for more than 72 hours (before meeting inclusion criteria)
* Symptomatic or uncorrected congenital heart disease or a right to left intra-cardiac shunt
* Any underlying condition that is likely to impair spontaneous respiratory drive/ efforts (Eg: Brainstem dysfunction, neuromuscular paralysis)
* Underlying chronic diseases (Eg: Cystic fibrosis, Chronic lung disease, etc)

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Twenty-eight-day ventilator-free days | 28 days

SECONDARY OUTCOMES:
Twenty-eight-day survival | 28 days
Length of PICU stay | Up to 3 months
  The children would be followed up for the duration of their PICU stay
Organ-failure-free-days | 28 days
Time-to-recovery of lung injury | Up to 28 days
  Number of days for recovery of lung injury (OI<5).
Number of children with adverse events | 3 years
  Children would be observed for incidence of adverse events during the period of PICU stay/ ventilation
All-cause mortality | Three months
Spirometry | 3 months
  Forced Expiratory volume during 1st second/ Forced vital capacity
Pediatric Cerebral performance category | 6 Months
  Functional outcomes
Pediatric Overall performance category | 6 months
Spirometry | 6 months
  Forced Expiratory Volume during 1st second / Forced Vital Capacity
Pediatric overall performance category | 3 months
  Assessment of functional outcomes
Pediatric cerebral performance category | 3 months
  Assessment of functional outcomes
Interleukin-6 levels | 72 hours of enrolment
Arterial lactate levels | 72 hours
Percentage reduction in 'oxygenation Index' | 6 hours
  Percentage improvement in oxygenation index at 6 hours of enrolment
Radiological score | 48 hours
Duration of inotropic requirement | up to 7 days
  Average time frame
Vaso-active inotropic score | 72 hours
Cumulative dose of sedation | 7 days
Cumulative dose of analgesic | 7 days
Cumulative dose of neuromuscular blocking agent | 7 days
Requirement for renal replacement therapy | 28 days
  Need for renal replacement therapy in the first 28 days of PICu stay or discharge/ death whichever is earlier
Pediatric Logistic Organ Dysfunction (PELOD) score | 7 days

OTHER OUTCOMES:
Recruitment rate | 3 years
  Number of children recruited per month on an average
Rate of enrolment among eligible children | 3 years
  Feasibility outcome Number of children who get enrolled in the study after consent among all eligible children
Contamination rate | 3 years
  Proportion of recruited children who cross-over from one arm to another
Attrition rate | 3 months
  Proportion of children who are lost to follow-up at 3 months
Protocol adherence rate | 3 years
  Proportion of children where all supportive care protocols are adhered to.

CONTACTS AND LOCATIONS:
Overall Officials: Saptharishi L G, MBBS, MD, Principal Investigator — DM (Pediatric Critical Care) Senior Resident, Division of Pediatric critical care, Dept Of Pediatrics, Advanced Pediatrics Center, PGIMER, Chandigarh, INDIA; Jayashree Muralidharan, MBBS, MD, Study Chair — Additional Professor, Division of Pediatric critical care, Dept of Pediatrics, Advanced Pediatrics Center, PGIMER, Chandigarh, India; Sunit C Singhi, MBBS, MD, Study Director — Chief, Division of Pediatric Critical Care, Professor & Head, Department of Pediatrics, Advanced Pediatrics Center, PGIMER, Chandigarh, India; Arun Bansal, MBBS, MD, Study Chair — Assistant Professor, Division of Pediatric Critical care, Dept of Pediatrics, Advanced Pediatrics Center, PGIMER, Chandigarh, India
Locations (1):
- Pediatric Intensive care unit, Division of Pediatric Critical Care, Advanced Pediatrics Center, Post-graduate Institute of Medical Education & Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided
Permission would have to be sought from institution in this regard.

REFERENCES:
- [Background] Andrews P, Habashi N. Airway pressure release ventilation. Curr Probl Surg. 2013 Oct;50(10):462-70. doi: 10.1067/j.cpsurg.2013.08.010. No abstract available. PMID 24156844
- [Background] Andrews PL, Shiber JR, Jaruga-Killeen E, Roy S, Sadowitz B, O'Toole RV, Gatto LA, Nieman GF, Scalea T, Habashi NM. Early application of airway pressure release ventilation may reduce mortality in high-risk trauma patients: a systematic review of observational trauma ARDS literature. J Trauma Acute Care Surg. 2013 Oct;75(4):635-41. doi: 10.1097/TA.0b013e31829d3504. PMID 24064877
- [Background] Emr B, Gatto LA, Roy S, Satalin J, Ghosh A, Snyder K, Andrews P, Habashi N, Marx W, Ge L, Wang G, Dean DA, Vodovotz Y, Nieman G. Airway pressure release ventilation prevents ventilator-induced lung injury in normal lungs. JAMA Surg. 2013 Nov;148(11):1005-12. doi: 10.1001/jamasurg.2013.3746. PMID 24026214
- [Background] Roy SK, Emr B, Sadowitz B, Gatto LA, Ghosh A, Satalin JM, Snyder KP, Ge L, Wang G, Marx W, Dean D, Andrews P, Singh A, Scalea T, Habashi N, Nieman GF. Preemptive application of airway pressure release ventilation prevents development of acute respiratory distress syndrome in a rat traumatic hemorrhagic shock model. Shock. 2013 Sep;40(3):210-6. doi: 10.1097/SHK.0b013e31829efb06. PMID 23799354
- [Background] Roy S, Habashi N, Sadowitz B, Andrews P, Ge L, Wang G, Roy P, Ghosh A, Kuhn M, Satalin J, Gatto LA, Lin X, Dean DA, Vodovotz Y, Nieman G. Early airway pressure release ventilation prevents ARDS-a novel preventive approach to lung injury. Shock. 2013 Jan;39(1):28-38. doi: 10.1097/SHK.0b013e31827b47bb. PMID 23247119
- [Derived] Lalgudi Ganesan S, Jayashree M, Chandra Singhi S, Bansal A. Airway Pressure Release Ventilation in Pediatric Acute Respiratory Distress Syndrome. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2018 Nov 1;198(9):1199-1207. doi: 10.1164/rccm.201705-0989OC. PMID 29641221